CLINICAL TRIAL: NCT03838393
Title: Prognosis of Trigeminal Neuralgia When Enrolled in a Multidisciplinary Management Program - a Two-year Prospective Real-life Study
Brief Title: Prognosis of Trigeminal Neuralgia When Enrolled in a Multidisciplinary Management Program
Status: Completed | Type: Observational
Sponsor: Danish Headache Center (Other)
Responsible Party: Principal Investigator, Tone Heinskou, medical doctor, Danish Headache Center
Other Study IDs: H-1-2012-093
Record Dates: First submitted 2019-02-06; First posted 2019-02-12 (Actual); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Trigeminal Neuralgia
Keywords: multidisciplinary management; real-life study
MeSH Terms: conditions — Trigeminal Neuralgia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: multidisciplinary management — pharmacological and non.pharmacological treatment (specially trained nurses, psychologists and physiologists)

SUMMARY:
Background: Prognosis of medically treated trigeminal neuralgia patients is assumed to be poor, but the evidence is lacking. Thus, prospective real-life studies of medical management of trigeminal neuralgia are warranted.

Methods: Observational study. Patients were consecutively enrolled in a structured management program at a specialist centre for facial pain. Optimisation of medical treatment, physiotherapy, psychotherapy, and advice from trained nurses, were parts of the program. Medically intractable patients were referred for neurosurgery. Data-collection was prospective using standardised schemes and patient surveys. The aim was to describe the two-year outcome of medical treatment at the specialist centre. The primary outcome was a 50% reduction in the overall burden of pain according to a Numerical Rating Scale (NRS) after two years.

This study aimed to provide evidence concerning the real-life efficacy of medical management of trigeminal neuralgia (TN) when directed by specialists. The investigatgors hypothesised that the two-year prognosis in a group of medically managed TN patients enrolled in a structured multidisciplinary management program was favourable, defined as a 50 % reduction of the overall burden of pain over a two-year period

ELIGIBILITY:
Inclusion criteria:

1. recordings of the intensity of pain at enrolment of the programme (baseline recording),
2. a two-year assessment (end-point recording),
3. recording of effect and side-effects of drug treatment (at baseline and endpoint).

The exclusion criteria

1. initiation of medical treatment at the DHC before May 2012,
2. neurosurgical treatment of TN within the two-year follow-up
3. incomplete two-year follow-up

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The diagnostic criteria used in this study were the beta version of the 3rd edition of the International Classification of Headache Disorders (ICHD-3-beta). Until the publication of IHCD-3-beta, ICHD 2 criteria were used. According to the ICHD-3 classification, this study included patients with both idiopathic and classical TN; in this paper termed primary TNThe number of patients enrolled in the inclusion period determined the sample size.
Sampling Method: Non-Probability Sample
Enrollment: 186 (Actual)
Dates: Start 2012-05 (Actual); Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
change in overall burden of pain NRS over a two-year period | 2 years
  Defined as a good outcome, i.e number of patients who had a reduction of minimum 50% on the NRS two years after enrolment in the management program compared with baseline

SECONDARY OUTCOMES:
No changes of the overall burden of pain NRS over the two-year follow-up period | 2 years
  Defined as poor outcome, i.e number of patients who had a no reduction the NRS two years after enrolment in the management program compared with baseline

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Heinskou TB, Maarbjerg S, Wolfram F, Rochat P, Brennum J, Olesen J, Bendtsen L. Favourable prognosis of trigeminal neuralgia when enrolled in a multidisciplinary management program - a two-year prospective real-life study. J Headache Pain. 2019 Mar 4;20(1):23. doi: 10.1186/s10194-019-0973-4. PMID 30832577